CLINICAL TRIAL: NCT06141200
Title: Efficacy and Safety of Roselle in Patients With Grade 1 Essential Hypertension: A Phase III, Randomized, Double-Blind, Double-Dummy, Active-Controlled Clinical Trial
Brief Title: NW Roselle in Grade 1 Essential Hypertension: Phase III Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Natural Wellness Egypt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-ROSELLE-572023
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Essential Hypertension
Keywords: Grade 1 Hypertension; primary hypertension; hibiscus; olive leaves; medicinal plants; blood pressure
MeSH Terms: conditions — Essential Hypertension | interventions — Captopril

STUDY DESIGN:
Intervention Model Description: A Phase III, Randomized, Parallel, Double-Dummy, Active-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Arm 1) (Experimental): The patient will receive NW Roselle capsules 1000 mg and placebo tablets. Patients will take two capsules of NW Roselle and one placebo tablet orally BID on an empty stomach with plenty of water 15 minutes before meals or one hour after meals.
  A total dose of 2000 mg of NW Roselle will be administered per day.
  Interventions: Drug: NW Roselle
- Control Group (Arm 2) (Active Comparator): Captopril 25 mg tablets will be used. The patient will receive placebo capsules and Captopril 25 mg tablets. Patients will take two placebo capsules and one Captopril 25 mg tablet orally BID on an empty stomach with plenty of water 15 minutes before meals or one hour after meals.
  A total dose of 50 mg of Captopril will be administered per day.
  Interventions: Drug: Captopril 25Mg Tab

INTERVENTIONS:
Drug: NW Roselle — NW Roselle is a powdered extract from the flowers of Hibiscus Sabdariffa (300mg) and the leaves of Olea europaea (200 mg).
  Arms: Study Group (Arm 1)
Drug: Captopril 25Mg Tab — Active Comparator
  Arms: Control Group (Arm 2)

SUMMARY:
In this Phase III clinical trial, researchers evaluate the efficacy and safety of NW Roselle®, a powdered medicinal product developed by Natural Wellness. NW Roselle combines extracts from Hibiscus Sabdariffa (HS) flowers and Olea europaea (OE) leaves. The trial aims to gather evidence on the efficacy and safety of NW Roselle as a potential treatment option for Grade 1 essential hypertension.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for heart, brain, and kidney diseases, and is a leading cause of death and illness globally. Natural Wellness has developed NW Roselle®, a powdered medicinal product that combines extracts from Hibiscus Sabdariffa (HS) flowers and Olea europaea (OE) leaves.

In this Phase III clinical trial, researchers are evaluating the efficacy and safety of NW Roselle, in the treatment of Grade 1 essential hypertension. Eligible participants who meet the criteria will be enrolled and randomized in a 1:1 ratio. They will be assigned to receive either NW Roselle or an active control, Captopril 25 mg twice daily.

Before the treatment begins, participants will provide informed consent and undergo assessments to collect information about their medical history, hypertension status, lifestyle factors, and demographics. Throughout the trial, the participant's vital signs, physical exams, and laboratory tests will be conducted to monitor their health and response to the treatment. Adherence to the assigned treatment will be monitored, and any potential adverse events or side effects will be tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with grade 1 essential hypertension (Systolic Blood Pressure: 140-159 mmHg, and/or Diastolic Blood Pressure 90-99 mmHg) (Williams et al., 2018).
2. Not currently taking any medication for hypertension.
3. Able and willing to provide written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with BMI > 45 Kg/m2 or BMI < 18 Kg/m2.
3. Patients with a known history of secondary hypertension (e.g., hyperaldosteronism, pheochromocytoma, renal artery stenosis, Cushing syndrome).
4. Renal impairment (Estimated Creatinine Clearance (Cr.Cl.) < 30 ml/min as measured by the Cockcroft-Gault formula).
5. Known Severe hepatic impairment, biliary cirrhosis, or cholestasis.
6. Patients with a history of arrhythmias, ischemic heart diseases, obstruction of the outflow tract of the left ventricle (e.g., hypertrophic obstructive cardiomyopathy, and high-grade aortic stenosis), congestive heart failure, valvular disease, myocardial infarction (MI), angina, myocardial revascularization, or cerebrovascular accident (CVA) within 6 months prior to study entry.
7. Participation in other clinical studies within 30 days before screening.
8. Known or suspected allergy or any contraindications to the trial products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The mean systolic blood pressure | Week 12
  The mean systolic blood pressure difference between the study arm and the control arm adjusted for baseline blood pressure.
The mean diastolic blood pressure | Week 12
  The mean diastolic blood pressure difference between the study arm and the control arm adjusted for baseline blood pressure.

SECONDARY OUTCOMES:
Systolic Blood Pressure Paired Change | Week 12
  The mean changes in systolic blood pressure between baseline and week 12 within each arm.
Diastolic Blood Pressure Paired Change | Week 12
  The mean changes in diastolic blood pressure between baseline and week 12 within each arm.
The rate of achieving blood pressure levels of (Systolic < 140 and Diastolic < 90 mmHg) by week 12 | Week 12
  The proportion of patients in each treatment group who are able to achieve the target blood pressure levels of systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg by week 12.
The rate of achieving systolic blood pressure range (120-130 mmHg) by week 12 | Week 12
  The proportion of patients in each treatment group who are able to achieve the target systolic blood pressure range of 120-130 mmHg by week 12.
The rate of achieving diastolic blood pressure range (70 - 80 mmHg) by week 12 | Week 12
  The proportion of patients in each treatment group who are able to achieve the target diastolic blood pressure control of 70-80 mmHg by week 12.
Compliance Rate | 12 weeks
  The mean medication compliance rate (%) will be calculated for each subject as: [(Total number of administered doses) / (Expected number of doses)] *100%.
Adverse events rate | 12 weeks
  2. The incidence of AEs reported by the patients, summarized by system organ class, severity, and relationship to study intervention, over the course of treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elkafrawy N, Younes K, Naguib A, Badr H, Kamal Zewain S, Kamel M, Raoof GFA, M El-Desoky A, Mohamed S. Antihypertensive efficacy and safety of a standardized herbal medicinal product of Hibiscus sabdariffa and Olea europaea extracts (NW Roselle): A phase-II, randomized, double-blind, captopril-controlled clinical trial. Phytother Res. 2020 Dec;34(12):3379-3387. doi: 10.1002/ptr.6792. Epub 2020 Jul 29. PMID 32725873
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in hypertension prevalence and progress in treatment and control from 1990 to 2019: a pooled analysis of 1201 population-representative studies with 104 million participants. Lancet. 2021 Sep 11;398(10304):957-980. doi: 10.1016/S0140-6736(21)01330-1. Epub 2021 Aug 24. PMID 34450083
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Background] Kandzari DE, Mahfoud F, Weber MA, Townsend R, Parati G, Fisher NDL, Lobo MD, Bloch M, Bohm M, Sharp ASP, Schmieder RE, Azizi M, Schlaich MP, Papademetriou V, Kirtane AJ, Daemen J, Pathak A, Ukena C, Lurz P, Grassi G, Myers M, Finn AV, Morice MC, Mehran R, Juni P, Stone GW, Krucoff MW, Whelton PK, Tsioufis K, Cutlip DE, Spitzer E. Clinical Trial Design Principles and Outcomes Definitions for Device-Based Therapies for Hypertension: A Consensus Document From the Hypertension Academic Research Consortium. Circulation. 2022 Mar 15;145(11):847-863. doi: 10.1161/CIRCULATIONAHA.121.057687. Epub 2022 Mar 14. PMID 35286164
- [Background] Abdel-Rahman RF, Hessin AF, Abdelbaset M, Ogaly HA, Abd-Elsalam RM, Hassan SM. Antihypertensive Effects of Roselle-Olive Combination in L-NAME-Induced Hypertensive Rats. Oxid Med Cell Longev. 2017;2017:9460653. doi: 10.1155/2017/9460653. Epub 2017 Oct 22. PMID 29201276